CLINICAL TRIAL: NCT00496925
Title: Examining the Usage of Dopamine Blockers in OCD Patients
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Chaim Sheba Medical Center
Other Study IDs: SHEBA- 07-4651-JZ-CTIL
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
We examine the usage of Dopamine blockers in OCD patients. We want to examine their frequency of usage, compare the course of the disease between those who receive and those who do not receive Dopamine blockers, and efficacy of the treatment.

The study will be done in two stages: 1. Collecting information the usage of Dopamine blockers from 150 OCD patients' files. 2. interviewing 60-70 patients to see the difference those who receive and those who do not receive Dopamine blockers in their current severity of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* DSM-IV diagnosis of OCD
* Ability to understand patient information sheet, and consent to participate

Exclusion Criteria:

* Current or past Psychotic or Bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient and Inpatients
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel